CLINICAL TRIAL: NCT05022979
Title: Prevalence of Micro-nutritional Deficiencies in Pregnant Women Presenting to the Emergency Department for Threatened Delivery
Brief Title: Prevalence and Risk Factors for Micronutrient Deficiencies During Pregnancy in Cayenne, French Guiana
Acronym: CarMa
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: CarMa
Record Dates: First submitted 2021-07-06; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Deficiency; Diet; Pregnancy
Keywords: micronutrients; risks factors; social inequalities
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational only — The investigator collected the patient's data from the medical record and interviewed the patient to complete the nutritional questionnaire.
  The required biological, blood and urine samples were collected during routine blood sampling upon entry and hospitalization.

SUMMARY:
Micronutrient deficiencies are frequent in pregnant women in French Guiana, a French territory in South America. Micronutrient deficiencies are more frequent in precarious women. Obesity is a frequent problem but it is also associated with micronutrient deficiency. Micronutrient deficiencies have largely been overlooked in this outermost European region and should be corrected.

DETAILED DESCRIPTION:
Involved in physical and brain development, immunity and metabolism, micronutrients have profound health effects. The nutritional status of pregnant women is a major determinant of fetal health. French Guiana has a rapid population growth. Social inequalities, cultural practices and gastrointestinal nematode infections in French Guiana could affect the prevalence of these deficiencies. The main objective of the present study was to estimate the prevalence of micronutrient deficiency among pregnant women in French Guiana. The secondary objective was to identify socio-demographic, dietary, obstetrical and neonatal risk factors associated with deficiencies.

Pregnant women over 22 weeks of pregnancy hospitalized for delivery at the Obstetrical Emergency Department of the Hospital Center in Cayenne from May 2018 to March 2019 were included. A socio-demographic and food questionnaire was administered. Medical data were collected from the medical records. Blood and urine samples were taken. The descriptive analysis used Student and Chi2 tests.

A total of 341 women were included. The majority were born in Haiti (39%) and French Guiana (34%). At least one micronutrient deficiency was observed in 81% of women. Precarious women had a significantly greater risk of micronutrient deficiency during pregnancy compared to those with both normal and complementary health insurance.

Micronutrient deficiencies in pregnant women in French Guiana are a public health problem, a fact that was previously overlooked in a context of rising obesity. With over half of women overweight or obese and 81% with at least 1 micronutrient deficiency, balanced nutrition should be a major focus.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at least 22 weeks of amenorrhea (WHO threshold for fetal viability)
* Patient hospitalized for delivery in the Gynecological and Obstetrical Emergency Unit at Cayenne hospital
* Patient's consent
* Consent of the legal representative if the patient is a minor

Exclusion Criteria:

* Refusalto participate in the study.
* Being under guardianship or curatorship
* Having been previously enrolled in the study

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any woman who was pregnant (22 weeks and more), hospitalized for delivery in the Gynecological and Obstetrical Emergency Unit at Cayenne hospital could participate in the studyafter giving written informed consent.The mode of delivery or urgent/non-urgent context did not influence the eligibility for inclusion. The criteria for non-inclusion were refusal to participate in the study; being under guardianship; and having already been enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Identification of a micronutrient deficiency defined as at least one micronutrient below the lower limit. | 1 day
  * urinary iodine < 100 µg/L
  * blood zinc level < 70 µg/dL
  * magnesium < 0.75 mmol/L
  * serum retinol < 0.70 µmol/L
  * erythrocyte folate < 305 nmol/L
  * blood cobalamin level < 150 pmol/L
  * Martial status: ferritin < 20 µg/L; serum iron < 15 µg/L; iron saturation coefficient of transferrin < 16%.

SECONDARY OUTCOMES:
Sociodemographic information | 1 day
  Socio-demographic and dietary risk factors associated with micronutrient deficiencies were investigated using a structured questionnaire.
assessment of Food diversity score | 1 day
  The food diversity score was inspired by the Food and Agriculture Organization's reports was assessed through a 24h recall, and calculated by adding the number of unique food groups consumed during last 24 hours.
Obstetrical and neonatal outcomes | 1 day
  Obstetrical and neonatal pathologies associated with micronutrient deficiencies were studied throughpatient interrogation and by analyzing medical records: rate of preeclampsia
Newborn health status | 1 day
  Gestational age at delivery, mode of delivery, weight, height, height, head circumference, APGAR, pathologies diagnosed on clinical examination before the 8th day of life
Mother Health status | 1 day
  Weight before pregnancy and on the day of inclusion, height, gestational age, pregnancy follow-up, microcytic anemia (hemoglobinemia <110 g/L, GMV >80 fl), primary hypothyroidism (increased TSH), gynaecological-obstetrical history, personal history of goiter or dysthyroidism, history of night blindness, personal history of anemia, other chronic conditions, history of digestive disorder/parasitoses, malaria history, drug treatment before and during pregnancy, micronutrient supplementation before and during pregnancy, tobacco use during pregnancy, alcohol use during pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duclau A, Abad F, Adenis A, Sabbah N, Leneuve M, Nacher M. Prevalence and risk factors for micronutrient deficiencies during pregnancy in Cayenne, French Guiana. Food Nutr Res. 2021 Feb 22;65. doi: 10.29219/fnr.v65.5268. eCollection 2021. PMID 33776616